CLINICAL TRIAL: NCT03575039
Title: The VITALE Study Evaluating Safety and Effectiveness/Performance of the Microport CardioFlow VitaFlow II - Transcatheter Aortic Valve System
Brief Title: VitaFlowTM II Transcatheter Aortic Valve System Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai MicroPort CardioFlow Medtech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Valve-2018-01
Record Dates: First submitted 2018-05-31; First posted 2018-07-02 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm clinical investigation (Experimental): Subjects in experimental group will be implanted the VitaFlow II Transcatheter Aortic Valve System.
  Interventions: Device: VitaFlow II Transcatheter Aortic Valve System

INTERVENTIONS:
Device: VitaFlow II Transcatheter Aortic Valve System — VitaFlow II Transcatheter Aortic Valve System contains a Valve stent -VitaFlow Aortic Valve, a Delivery system-VitaFlow II Delivery System and a Introducer set

SUMMARY:
A prospective, single arm clinical investigation evaluating safety and effectiveness/performance of the Microport CardioFlow VitaFlowTM II - Transcatheter Aortic Valve System for the treatment of symptomatic severe aortic stenosis via transcatheter access in increased surgical risk patients

DETAILED DESCRIPTION:
This is a prospective, multicenter, single arm and controlled clinical investigation compared to recent historical results. The purpose is to evaluate the safety, performance and efficacy of the VitaflowTM II Transcatheter Aortic Valve system.

The entire system including valve system, delivery system and introducer system. We will implant the valve system into subjects and followed up them for 5 years after the procedure. This clinical trial will be conducted in 15 sites in Europe.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of age > 18 years
2. Subjects suffering from severe aortic valve stenosis, including bicuspid and tricuspid valves, defined as follows:

   High-gradient aortic stenosis (mean pressure gradient across aortic valve >40 mmHg or peak velocity ≥4.0 m/s.
3. Subject has symptomatic valve stenosis presenting with NYHA ≥ Class II
4. Subjects with a documented heart team agreement of increased surgical risk as described in the population
5. ECG-gated multi-slice computed tomographic (MSCT) measurements determined an aortic annulus or supra-annular diameter ≥17 and ≤29mm. Findings of TTE, TEE and conventional aortography should be integrated in the anatomic assessment, when performed
6. Patient deemed eligible by Centralised Case Review Committee (CRC) assessment recommends VitaFlow™ II Transcatheter Aortic Valve System implantation
7. Subject can understand the purpose of the clinical investigation, has signed voluntary the informed consent form and is agreeing to the scheduled follow up requirements

Exclusion Criteria:

1. Arterial aorto-iliac-femoral axis unsuitable for transfemoral access as assessed by conventional angiography and/or multi-detector computed tomographic angiography (access vessel diameter incompatible with a 19 to 22F OD delivery system with integrated sheath or 21 to 24F OD sheath)
2. Aortic root anatomy condition or lesion preventing implantation or access to the aortic valve
3. Non-calcific acquired aortic stenosis
4. Native unicuspid aortic valve or congenital aortic abnormality (except for bicuspid aortic valve) not permitting TAVI
5. Previous implantation of heart valve in any position
6. Severe aortic regurgitation (>3+)
7. Severe mitral regurgitation (>3+)
8. Severe tricuspid regurgitation (>3+)
9. Severe left ventricular (LV) dysfunction (left ventricular ejection fraction < 30%)
10. Echocardiographic evidence of intracardiac mass, thrombus or vegetation
11. Multi-vessel coronary artery disease with a Syntax score or residual Syntax score > 22 and/or unprotected left main coronary artery.
12. Cardiogenic shock manifested by low cardiac output, vasopressor dependence, or mechanical hemodynamic support
13. Untreated cardiac conduction disease in need of pacemaker implantation
14. Uncontrolled atrial fibrillation (resting heart rate > 120bpm)
15. Active and/or suspicion of endocarditis or ongoing sepsis
16. Blood dyscrasias defined as: leukopenia (WBC<1000 mm3), thrombocytopenia (PLT<50,000 cells/mm3), history of bleeding diathesis or coagulopathy, or hypercoagulable states
17. Evidence of an acute myocardial infarction ≤ 1 month (30 days) before signing informed consent
18. Any need for emergency surgery
19. Recent (within 6 months of signing informed consent) cerebrovascular accident (CVA) or transient ischemic attack (TIA)
20. Symptomatic carotid or vertebral artery disease or successful treatment of carotid stenosis within 30 days prior to signing informed consent
21. Any active bleeding that precludes anticoagulation
22. Liver failure (Child-C)
23. End-stage renal disease requiring chronic dialysis or creatinine clearance < 20cc/min
24. Pulmonary hypertension (systolic pressure >80mmHg)
25. Severe chronic pulmonary disease (COPD) demonstrated by an expiratory volume (FEV1) < 750cc
26. Refusal of blood transfusion
27. A known hypersensitivity or contraindication to all anticoagulation/antiplatelet regimens (or inability to be anticoagulated for the index procedure), to nitinol, to dairy products, to polyethylene terephthalate (PET) or contrast media
28. Any medical, social or psychological condition that in the opinion of the investigator precludes the subject from giving appropriate consent or adherence to the required follow up procedures
29. Currently participating in another drug or device trial (excluding registries) for which the primary endpoint has not been assessed
30. Estimated life expectancy of less than 12 months
31. For female - pregnancy or intention to become pregnant prior to completion of all follow up procedures
32. Inability to comply with the clinical investigation follow-up or other clinical investigation requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Rate of all-cause mortality at 12 months post implantation | 12 months post implantation
  all-cause mortality including cardiovascular and non-cardiovascular

SECONDARY OUTCOMES:
Rate of Composite of all-cause mortality and disabling stroke | at 30 days, 6 months,12 months, 2, 3, 4 and 5 years post implantation
  defined as the ratio of all-cause dead and disabled subjects to total subjects at each time point
Rate of stroke (disabling and non-disabling) | at 30 days, 6 months,12 months, 2, 3, 4 and 5 years post-implantation
  defined as the ratio of stroke subjects (disabling and non-disabling) to total subjects at each time point
Initial success | within 30 days post-implantation
  defined as absence of procedural mortality AND correct positioning of a single VitaFlowTM Aortic Valve into the proper anatomical location AND absence of patient / VitaFlowTM Aortic Valve mismatch AND mean aortic valve gradient less than (<) 20 mmHg or peak velocity less than (<) 3m/s, AND absence of moderate or severe prosthetic valve regurgitation
Recapture success rate (when attempted) | at 1st day post-implantation
  defined as VitaFlowTM Aortic Valve is fully re-sheathed into the VitaFlowTM II delivery system, as verified by fluoroscopy
Successful insertion | at 1st day post-implantation
  navigation and functioning of ALL features for the VitaFlowTM II delivery system, deployment and implantation of the VitaFlowTM aortic valve and subsequent retrieval of the VitaFlowTM II delivery system
Valve function | at 30 days, 6 and 12 months and 2, 3, 4, 5 years post-implantation
  Evaluating valva function(including valve position, morphology, function and rate of valvular stenosis, valve regurgitation, orifice area and pressure gradient and paravalvular leakage) at each time point.
Changes in quality of life KCCQ | at 30 days, 6 and 12 months and 2, 3, 4, 5 years post-implantation compared to baseline
  an overall summary score can be derived from the physical function, symptom (frequency and severity), social function and quality of life domains. For each domain, the validity, reproducibility, responsiveness and interpretability have been independently established. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Changes in quality of life EQ-5D-5L | at 30 days, 6 and 12 months and 2, 3, 4, 5 years post-implantation compared to baseline
  Use the questions and score system to evaluate life quality of subjects at each The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Changes in frailty (KATZ questionnaire) | at 30 days, 12 months, 1, 2, 3, 4 and 5 years post-implantation compared to baseline
  Assesses the ability of patients to conduct activities of daily living by questions in KATZ questionnaire. We use dependent(0 points) and independent(1 points) to evaluate bathing, dressing, toileting, transferring, contience and feeding activities of subjects. Total score is 6 points, the higher the score, the more indepent of subjects.
Changes in cardiac function | at discharge, 30 days, 6 and 12 months and 2, 3, 4, 5 years post-implantation
  defined as changes in cardiac function at each time point according to the NYHA Classification Scheme compared to baseline
Rate of all-cause mortality | at 30 days, 6 months and 2, 3, 4, 5 years post-implantation
  all-cause mortality including cardiovascular and non-cardiovascular
Rate of main adverse cardiac and cerebral events (MACCE) | at 30 days, 6 and 12 months and 2, 3, 4, 5 years post-implantation
  Rate of main adverse cardiac and cerebral events (MACCE) including disabling stroke, myocardial infarction, open surgery, and new permanent pacemaker at each time point
Rate of life-threatening, disabling or severe bleeding (BARC 3 to 5) | at 30 days, 6 and 12 months and 2, 3, 4, 5 years post-implantation
  BARC 3 to 5 defined as in BARC definition in annex of the protocol
Rate of acute kidney injury network stage 2 and 3 or renal alternation therapy | at 30 days, 6 and 12 months and 2 to 5 years
  renal alternation therapy including haemodialysis, peritoneal dialysis and hemofiltration
Rate of implant related new and/or worsened conduction disturbances and arrhythmias, and occurrence of new permanent pacemaker implantation | at 30 days, 6 and 12 months and 2, 3, 4, 5 years post-implantation
  Rate of implant related new and/or worsened conduction disturbances and arrhythmias, and occurrence of new permanent pacemaker implantation
Rate of major vascular complications | at 30 days, 6 and 12 months and 2, 3, 4, 5 years post-implantation
  vascular complications defined according to VARC2 definitions
Rate of the occurrence of hospitalization | at 6, 12 months, and 2, 3, 4, 5 years post-implantation
  Rate of the occurrence of hospitalization for valve-related symptoms or worsening congestive heart failure
Rate of other TAVI-related adverse events | at 30 days, 6 and 12 months and at 2, 3, 4 and 5 years post implantation.
  Rate of other TAVI-related adverse events (conversion to open surgery, unplanned used of cardiopulmonary bypass, coronary obstruction requiring intervention, ventricular septal perforation, mitral valve apparatus damage or dysfunction, cardiac tamponade, endocarditis, valve thrombosis, valve mal-positioning, TAV-in-TAV deployment, structural valve deterioration, valve related dysfunction or events requiring repeat procedure [BAV, TAVR, SAVR]

CONTACTS AND LOCATIONS:
Overall Officials: Nicolo Piazza, Principal Investigator — Bern Unversity Hospital

IPD SHARING:
Plan to Share IPD: No
This is an internal clinical research, the detail data won't be shared with other researcher before our product come into the market.